CLINICAL TRIAL: NCT05216770
Title: Understanding Disorder-specific Neural Pathophysiology in Laryngeal Dystonia and Voice Tremor
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Kristina Simonyan, Professor of Otolaryngology - Head and Neck Surgery, Massachusetts Eye and Ear Infirmary
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2021P003142
Record Dates: First submitted 2021-11-27; First posted 2022-02-01 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Laryngeal Dystonia; Spasmodic Dysphonia; Tremor
MeSH Terms: conditions — Dysphonia; Tremor | interventions — Neuroimaging; Bupivacaine

STUDY DESIGN:
Intervention Model Description: Only one of three arms includes Intervention. The other two arms are Observational. The Interventional arm has a parallel study model where patients with laryngeal dystonia and voice tremor will be assigned to laryngeal sensory block in parallel. Allocation will be non-randomized.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Spatial and temporal CNS pathophysiology of laryngeal dystonia and voice tremor (Other): Simultaneous fMRI with EEG and MEG imaging will be used to examine neural dynamics during phonation.
  Interventions: Other: Brain imaging
- Sensorimotor modulations of laryngeal dystonia and voice tremor with bupivacaine (Active Comparator): Topical laryngeal block (1 ml of 0.75% bupivacaine solution) will be used to modulate somatosensory feedback from the laryngeal mucosa during speech production and examine associated changes in brain activity.
  Interventions: Drug: Laryngeal sensory block with topical bupivacaine
- Motor learning and CNS pathophysiology of laryngeal dystonia and voice tremor (Other): Implicit learning of the production of motor sequences will be examined during simultaneous fMRI/EEG and MEG imaging.
  Sensorimotor adaptation of speech production during MEG imaging will be examined during perturbing pitch or formants of auditory feedback consistently during speech production and examining the behavioral and neural correlates of the resulting across-trial adaptation responses.
  Interventions: Other: Brain imaging
- Placebo effects in laryngeal dystonia and voice tremor (Placebo Comparator): 1 ml of saline placebo matching to 1 ml of 0.75% bupivacaine solution will be used for a comparison with the topical laryngeal block to modulate somatosensory feedback from the laryngeal mucosa during speech production and examine associated changes in brain activity.
- Auditory feedback processing in laryngeal dystonia and voice tremor (Other): The role of auditory feedback processing on task-induced speech sensorimotor activity will be examined using MEG imaging during perturbing pitch or formants of auditory feedback, unpredictably during speech production, and examining the behavioral and neural correlates of the resulting within-trial compensation responses.
  Interventions: Other: Brain imaging

INTERVENTIONS:
Other: Brain imaging — Brain images will be conducted with function MRI, magnetoencephalography (MEG), and electroencephalography (EEG) to identify disorder-specific neural markers
  Arms: Auditory feedback processing in laryngeal dystonia and voice tremor; Motor learning and CNS pathophysiology of laryngeal dystonia and voice tremor; Spatial and temporal CNS pathophysiology of laryngeal dystonia and voice tremor
Drug: Laryngeal sensory block with topical bupivacaine — Laryngeal sensory block with bupivacaine will be used to modulate sensory feedback from vocal fold mucosa and examine the impact of sensory feedback on abnormal neural activity in LD and VT
  Arms: Sensorimotor modulations of laryngeal dystonia and voice tremor with bupivacaine

SUMMARY:
The researchers will examine functional neural correlates that differentiate between laryngeal dystonia and voice tremor and contribute to disorder-specific pathophysiology using a cross-disciplinary approach of multimodal brain imaging.

DETAILED DESCRIPTION:
Laryngeal dysphonia (LD) and Voice Tremor (VT) are neurological voice disorders that impair speech production. The characteristic feature of LD (i.e., occurring during speaking but not laughing or crying) and the lack of physical laryngeal abnormalities suggests that LD is likely a disorder affecting the task-specific control of phonation by the central nervous system (CNS). Similarly, VT is often observed without any clear peripheral laryngeal etiology, also suggesting a central origin but distinct from that affected in LD. The overall goal of this project is to characterize the common and distinct features of CNS pathophysiology in the neurological voice disorders, LD and VT. The act of speech is a dynamic process, including initial glottal movement, voice onset, and compensatory responses to sensory feedback fluctuations during sustained phonation. Identifying specific functional impairments in LD and VT requires a clear understanding of when in the process of phonation, as well as where in the CNS, aberrant activity occurs. Due to their poor temporal resolution, prior neuroimaging studies have not been able to address the question of when abnormal CNS activation occurs relative to specific phonation events. As a result, critical clues about the underlying etiologies in these disorders have likely been missed. A multimodal brain imaging will asses CNS abnormalities associated with LD and VT, specifically 1) Spatial and temporal CNS pathophysiology during speech and other vocal tasks; 2) Sensorimotor modulations on CNS pathophysiology; and 3) Motor learning and CNS pathophysiology. Future treatments for LD and VT can be developed by targeting CNS pathophysiological mechanisms identified in this project.

ELIGIBILITY:
Inclusion criteria:

1. Males and females of diverse racial and ethnic background;
2. Age 18-80 years;
3. Native English speakers;
4. Right-handed;
5. Normal cognitive status;
6. Patients will have laryngeal dystonia or voice tremor;
7. Healthy controls will be healthy individuals without neurological, psychiatric or otolaryngological problems.

Exclusion criteria:

1. Subjects who are incapable of giving informed consent;
2. Pregnant or breastfeeding women until a time when they are no longer pregnant or breastfeeding. All women of childbearing potential will have a urine pregnancy test performed before MRI, which must be negative for participation in the imaging studies;
3. Subjects with a past or present medical history of (a) neurological problems, such as stroke, movement disorders (other than specified LD and VT in the patient groups), brain tumors, traumatic brain injury with loss of consciousness, ataxias, myopathies, myasthenia gravis, demyelinating diseases; (b) psychiatric problems, such as schizophrenia, bipolar depression, obsessive-compulsive disorder, alcoholism, drug dependence; (c) laryngeal problems, such as vocal fold paralysis, paresis, vocal fold nodules and polyps, carcinoma, chronic laryngitis;
4. Patients with any other form of dystonia;
5. Patients who have dystonia symptoms at rest or have a presence of mirror dystonia;
6. Patients who are not symptomatic due to treatment with botulinum toxin injections into the affected muscles. The duration of positive effects of botulinum toxin varies from patient to patient but lasts, on average, for 3-4 months. All patients will be evaluated to ensure that they are fully symptomatic and are at least 3 months post-injection before participation;
7. To avoid the confounding effect of centrally acting drugs, all study participants will be questioned about any prescribed or over-the-counter medications as part of their initial screening. Those patients who receive medication(s) affecting the central nervous system will be excluded;
8. Patients will be asked whether they have undergone any head or neck surgery, which resulted in changes in regional anatomy or innervation. Because brain or laryngeal surgery may potentially lead to brain structure and function re-organization, all patients with such a history will be excluded;
9. Subjects who have certain tattoos and ferromagnetic objects in their bodies (e.g., implanted stimulators, surgical clips, prosthesis, artificial heart valve) that cannot be removed for MRI studies.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2022-03-24 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Functional MRI, MEG and EEG signal changes in laryngeal dystonia compared to voice tremor | 5 years
  Qualitative analysis of brain regions with disorder-specific increases and decreases of spatial (functional MRI) and temporal (MEG and EEG) signals will be determined in patients with laryngeal dystonia compared to patients with voice tremor
Effects of sensorimotor brain modulation on voice function in laryngeal dystonia | 5 years
  Quantitative measures of symptoms will be determined using Burk-Fahn-Marsden Dystonia Rating Scale where higher score means a worse outcome, following sensorimotor feedback modulation in patients with laryngeal dystonia
Effects of sensorimotor brain modulation on voice function in voice tremor | 5 years
  Quantitative measures of symptoms will be determined using Fahn-Tolosa-Marin Rating Scale where higher score means a worse outcome, following sensorimotor feedback modulation in patients with voice tremor

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Simonyan, MD, PhD, Study Director — Professor of Otolaryngology - Head and Neck Surgery
Locations (1):
- Massachusetts Eye and Ear and University of California San Francisco, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No